CLINICAL TRIAL: NCT03549156
Title: Comparison of a Two Ready-to-use Supplementary Foods of Differing Protein Quality for the Treatment of Moderate Acute Malnutrition in Rural Malawian Children: a Randomised, Investigator-blinded, Clinical Effectiveness Trial.
Brief Title: Comparison of a Two Ready-to-use Supplementary Foods of Differing Protein Quality for the Treatment of MAM.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Arla Foods (Industry); Kamuzu University of Health Sciences (Other); Project Peanut Butter (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 201805096
Record Dates: First submitted 2018-05-18; First posted 2018-06-07 (Actual); Last update posted 2020-03-16 (Actual); Status verified 2020-03

CONDITIONS: Malnutrition
Keywords: Moderate Acute Malnutrition, Malnutrition
MeSH Terms: conditions — Malnutrition

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Each food will be randomized to two colors with the study coordinator, nurse, caregivers blinded to the which color is which food.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- C-RUSF (Active Comparator): Control/Standard RUSF
  Interventions: Dietary Supplement: C-RUSF
- HIPRO RUSF (Active Comparator): New RUSF product
  Interventions: Dietary Supplement: HIPRO RUSF

INTERVENTIONS:
Dietary Supplement: C-RUSF — -RUSF contains whey permeate, WPC 80, peanut paste, sugar, soy oil, canola oil, a customized micronutrient premix to account for the minerals in whey permeate, and an emulsifier
  Other Names: Ready-to-use supplementary food
  Arms: C-RUSF
Dietary Supplement: HIPRO RUSF — HIPRO RUSF contains extruded soy flour, skimmed milk, peanut paste, sugar, soy oil, palm oil, a premix containing concentrated minerals and vitamins, an emulsifier and dicalcium phosphate or calcium carbonate
  Other Names: Ready-to-use supplementary food
  Arms: HIPRO RUSF

SUMMARY:
This is a prospective, randomised, double-blinded, controlled clinical effectiveness trial of two supplementary foods in the treatment of MAM. The setting will be 21 rural sites in southern Malawi. The participants will be 1800 children 6-59 months old with MAM, defined as mid-upper arm circumference (MUAC) ≥ 11.5 cm and < 12.5 cm and/or a weight-for-height Z-score (WHZ) between -2 and -3 without bipedal edema. Children will receive approximately 75 kcal/kg/d (314 kJ/kg/d) of one of two RUSFs in two-week rations for outpatient therapy of MAM. The two supplements will be a novel, locally produced peanut/dairy RUSFs, one with a high protein quality (HIPRO RUSF) or one with a standard protein quality, referred to as control RUSF (C-RUSF). The primary outcome measures will be recovery from MAM (achieving MUAC ≥ 12.5 cm and/or WHZ>-2 by 12 weeks) or failure (death, development of severe acute malnutrition, transfer to hospital for inpatient care, failure to recover from MAM by 12 weeks, default). Secondary outcome measures include rates of weight, height, and mid-upper-arm circumference (MUAC) gain, time to graduation, and adverse effects from the supplementary foods.

ELIGIBILITY:
Inclusion Criteria:

* MUAC < 12.5 cm and ≥ 11.5 cm
* without bipedal edema

Exclusion Criteria:

* simultaneously involved in another research trial or supplemental feeding program
* developmentally delayed, have a chronic debilitating illness such as cerebral palsy
* history of peanut or milk allergy

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 1858 (Actual)
Dates: Start 2018-06-25 (Actual); Primary Completion 2019-03-08 (Actual); Study Completion 2019-03-08 (Actual)

PRIMARY OUTCOMES:
Recovery from Moderate Acute Malnutrition using Mid-Upper Arm Circumference (MUAC) and Weight for Height Z score (WHZ) | 12 weeks
  Number of participants achieving a Mid-Upper Arm Circumference (MUAC) ≥ 12.5 cm and/or WHZ>-2 within a 12 week treatment period

CONTACTS AND LOCATIONS:
Overall Officials: Mark Manary, MD, Principal Investigator — Washington University School of Medicine in St. Louis
Locations (1):
- Local Feeding Clinics, Blantyre, Malawi